CLINICAL TRIAL: NCT00326001
Title: AURUM 8 - Ablation of the Cavotricuspid Isthmus in Patients With Atrial Flutter Using an 8 mm Gold Alloy Tip Electrode
Brief Title: Isthmus Ablation With Gold Electrode for Treatment of Atrial Flutter (AURUM 8)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP016
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2009-08

CONDITIONS: Atrial Flutter
Keywords: Transvenous Catheter Ablation; Radiofrequency Catheter Ablation; Atrial flutter; Catheter Ablation
MeSH Terms: conditions — Atrial Flutter

ARMS (2):
- Gold tip catheter (Experimental): Gold tip catheter
  Interventions: Device: Gold tip catheter
- Platinum-iridium tip catheter (Active Comparator): Platinum-iridium tip catheter
  Interventions: Device: Platinum-iridium tip catheter

INTERVENTIONS:
Device: Gold tip catheter — Radiofrquency ablation using gold tip catheter
  Arms: Gold tip catheter
Device: Platinum-iridium tip catheter — Radiofrequency ablation using platinum-iridium tip catheter
  Arms: Platinum-iridium tip catheter

SUMMARY:
The purpose of this study is to demonstrate the advantage of using a gold alloy tip electrode over a platinum/iridium alloy tip electrode in ablation of the cavotricuspid isthmus in patients with atrial flutter.

DETAILED DESCRIPTION:
Transvenous catheter ablation has become the therapy of choice for patients with recurring, isthmus-dependent right atrial flutter. Achieving bidirectional conduction block in the cavotricuspid isthmus is decisive for both acute and long-term therapy success and essentially depends on the selected ablation method and the lesion size. By using an 8 mm tip electrode instead of a conventional 4 mm electrode, deeper lesions can be made, thus significantly reducing the required number of energy applications for achieving a bidirectional conduction block. Experimental studies have proven that using an ablation electrode made of gold alloy allows the creation of deeper lesions than with conventional platinum-iridium electrodes. Due to the greater heat conductivity of the gold alloy as opposed to platinum-iridium, the cooling of the ablation electrode is improved and more electric energy can be transmitted to the tissue at identical temperatures.

The combination of both technologies in the form of an 8 mm-long gold electrode anticipates that the lesion depth required for an isthmus block can be achieved more quickly in comparison to the platinum-iridium electrode.

ELIGIBILITY:
Inclusion Criteria:

* At least one electrocardiogram (ECG)-documented (can be older than 3 months), symptomatic, typical atrial flutter episode with either negative, sawtooth-shaped P-waves in leads II, III, and augmented voltage foot (aVF), or positive P-waves in leads II, III, and aVF
* At least one persistent, typical atrial flutter episode of over 2 hours that has been documented in the history in the patient file and/or ECG
* Signed informed consent form

Exclusion Criteria:

* Patient has recently undergone isthmus ablation
* Acute coronary syndrome or myocardial infarction within the last 3 months
* Acute reversible causes for atrial flutter (e.g. acute myocarditis)
* Severe cardiac valvular defects
* Tricuspid valve replacement
* Atrial septum defect
* Cardiovascular surgery scheduled within the next 6 months
* Unstable medication in the last 7 days before study inclusion
* New York Heart Association (NYHA) class IV
* Women who are breastfeeding
* Pregnancy
* Abuse of drugs or alcohol
* Patient is unable to participate in follow-up examinations
* The patient has only partial legal competence
* Participation in another clinical study
* The ablation procedure presents an above average risk to the patient as compared to the normal patient group (must be noted by the physician on the appropriate form).
* Right atrial thrombus

Late Exclusion Criteria:

* Patient included by accident
* Premature termination of the ablation procedure
* Atrial flutter not dependent on the posterior isthmus
* No conduction at the posterior isthmus before ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Lewalter, Assoc. Prof. Dr., Principal Investigator — Universitätsklinikum Bonn, Medizinische Klinik and Poliklinik II, Sigmund-Freud-Strasse 25, D-53105 Bonn, Germany
Locations (28):
- Institute of Clinical and Experimental Medicine, Prague, Czechia
- Germany (24):
  - Universitätsklinik der RWTH Aachen, Aachen
  - Kerckhoff Klinik, Bad Nauheim
  - Charité Campus Mitte, Medizinische Fakultät der Humboldt Universität zu Berlin, Berlin
  - Vivantes Klinikum Am Urban, Berlin
  - Universitätsklinikum Charité, Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Charité, Campus Buch Franz-Volhard-Klinik, Berlin
  - Universitätsklinikum Charité, Campus Virchow-Klinikum, Berlin
  - Berufsgenossenschaftliche Kliniken, Bergmannsheil Universitätsklinik, Bochum
  - Medizinische Einrichtungen der Rheinischen Friedrich-Wilhelms-Universität Bonn, Bonn
  - Elektrophysiologische Praxis am Zentralkrankenhaus Links Der Weser, Bremen
  - Herzzentrum Duisburg, Duisburg
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Georg-August-Universität, Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Allgemeines Krankenhaus Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätskliniken des Saarlandes, Homburg/Saar
  - St. Vincentius Krankenhaus/St. Marien Krankenhaus - Abteilung für Innere Medizin III, Karlsruhe
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universitätsklinikum Mainz, Mainz
  - Städtisches Krankenhaus München-Bogenhausen, München
  - Universitätsklinikum Ulm, Ulm
  - Klinikum der Stadt Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Medizinische Universitätsklinik Würzburg, Würzburg
- Hungary (3):
  - Semmelweis Medical University - Department of Cardiology, Budapest
  - The Debrecen University of Medicine, Center of Medicine and Health Care Sciences, Clinical Department of Cardiology, Debrecen
  - The University of Pecs, Pécs

REFERENCES:
- [Background] Lewalter T, Bitzen A, Wurtz S, Blum R, Schlodder K, Yang A, Lickfett L, Schwab JO, Schrickel JW, Tiemann K, Linhart M, Zima E, Merkely B, Luderitz B. Gold-tip electrodes--a new "deep lesion" technology for catheter ablation? In vitro comparison of a gold alloy versus platinum-iridium tip electrode ablation catheter. J Cardiovasc Electrophysiol. 2005 Jul;16(7):770-2. doi: 10.1111/j.1540-8167.2005.40832.x. PMID 16050836
- [Background] Berjano EJ. Gold-tip electrodes--a new 'deep lesion' technology for catheter ablation? In vitro comparison of gold alloy versus platinum-iridium tip electrode ablation catheter. J Cardiovasc Electrophysiol. 2005 Dec;16(12):1395-6. doi: 10.1111/j.1540-8167.2005.280_2.x. No abstract available. PMID 16403084
- [Derived] Lickfett L, Mittmann-Braun E, Weiss C, Spencker S, Jung W, Haverkamp W, Willems S, Deneke T, Kautzner J, Wiedemann M, Siebels J, Pitschner HF, Hoffmann E, Hindricks G, Zabel M, Vester E, Schwacke H, Leyen JV, Mewis C, Bauer W, Lewalter T. Differences in clinical and echocardiographic parameters between paroxysmal and persistent atrial flutter in the AURUM 8 study: targets for prevention of persistent arrhythmia? Pacing Clin Electrophysiol. 2013 Feb;36(2):194-202. doi: 10.1111/pace.12051. PMID 23379836
- [Derived] Lewalter T, Weiss C, Spencker S, Jung W, Haverkamp W, Willems S, Deneke T, Kautzner J, Wiedemann M, Siebels J, Pitschner HF, Hoffmann E, Hindricks G, Zabel M, Vester E, Schwacke H, Mittmann-Braun E, Lickfett L, Hoffmeister S, Proff J, Mewis C, Bauer W; AURUM 8 Study Investigators. Gold vs. platinum-iridium tip catheter for cavotricuspid isthmus ablation: the AURUM 8 study. Europace. 2011 Jan;13(1):102-8. doi: 10.1093/europace/euq339. Epub 2010 Sep 28. PMID 20876601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 463 patients were enrolled in the AURUM 8 study from June 2004 to March 2007 in 19 clinical centers in Germany and the Czech Republic.
Pre-assignment Details: No exclusion before assignment
Groups:
- Gold Tip Catheter: Patients allocated to be ablated by 8-mm gold tip catheter
- Pt-Ir Tip Catheter: Patients allocated to be ablated by 8-mm Platinum-Iridium tip catheter
Period: Overall Study
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter
Started | 236 | 227
Completed | 229 | 219
Not Completed | 7 | 8
Not completed — Adverse Event | 4 | 5
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter | Total
Number analyzed (Participants) | 236 | 227 | 463
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 92 | 189
  >=65 years | 139 | 135 | 274
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 66 (11) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 80
  Male | 191 | 192 | 383
Region of Enrollment [Number; unit: participants]
  Czech Republic | 9 | 8 | 17
  Germany | 227 | 219 | 446

OUTCOME MEASURES:

1. Primary Outcome: Duration of Energy Application
Description: Cumulative amount of time current is flowing through the catheter tip. The current (in the radiofrequency range) is applied to ablate the cavotricuspid isthmus in the right atrium.
Time Frame: ablation procedure
Population: Per protocol
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter
Number analyzed (Participants) | 229 | 219
minute | 10.2 (6.9) | 10.9 (6.9)
Statistical Analysis 1: Comparison: Gold Tip Catheter vs Pt-Ir Tip Catheter; Test type: Superiority or Other; p = 0.25, t-test, 2 sided — P-value not adjusted for multiple comparisons

2. Secondary Outcome: Ablation Success With the First Catheter
Description: Delivery of radiofrequency current was repeated until a cavotricuspid isthmus (CTI) conduction block was detected. The final bidirectional CTI block test (well documented in the literature) was performed 20 minutes after the last radiofrequency current delivery to assess ablation success (Y/N).
  Positive final bidirectional cavotricuspid isthmus condution block test means "ablation successful".
  Negative final bidirectional cavotricuspid isthmus condution block test means "ablation unsuccessful"; ablation should be continued until success or terminated and classified as unsuccess.
Time Frame: ablation procedure
Population: per protocol
Measure: Number; unit: Patients
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter
Number analyzed (Participants) | 229 | 219
Patients | 216 | 195
Statistical Analysis 1: Comparison: Gold Tip Catheter vs Pt-Ir Tip Catheter; Test type: Superiority or Other; p = 0.042, Chi-squared

3. Secondary Outcome: Number of Patients With Long-term Treatment Success
Description: No recurrence of atrial flutter after ablation
Time Frame: 6 months after ablation
Population: per protocol
Measure: Number; unit: Patients
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter
Number analyzed (Participants) | 229 | 219
Patients | 225 | 213
Statistical Analysis 1: Comparison: Gold Tip Catheter vs Pt-Ir Tip Catheter; Test type: Superiority or Other; p = 0.53, Chi-squared

4. Secondary Outcome: Number of Patients With Charred Catheter Tips
Description: Char or coagulum formation on the catheter tip
Time Frame: ablation procedure
Population: per protocol
Measure: Number; unit: Patients
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter
Number analyzed (Participants) | 229 | 219
Patients | 11 | 83
Statistical Analysis 1: Comparison: Gold Tip Catheter vs Pt-Ir Tip Catheter; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Gold Tip Catheter | Pt-Ir Tip Catheter
Serious Adverse Events (participants affected / at risk) | 20/229 | 12/219
Other Adverse Events (participants affected / at risk) | 0/229 | 0/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gold Tip Catheter (N=229) | Pt-Ir Tip Catheter (N=219)
Death (General disorders) | 2 (2) | 1 (1) — Death for any cause
Hospitalization (General disorders) | 18 (18) | 12 (12) — Hospitalization for any cause

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No